CLINICAL TRIAL: NCT06265662
Title: A Digital Health Program for Non-Communicable Disease Prevention in a Workplace Setting in Thailand: A Quasi-Experimental Study
Brief Title: A Digital Health Program for Non-Communicable Disease Prevention in a Workplace Setting in Thailand
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Zethapong Nimmanterdwong, MD, Student, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 66701100301
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Chronic Disease; Noncommunicable Diseases
Keywords: Mobile Health; Self Care; Workplace; Health Promotion; Digital Medicine
MeSH Terms: conditions — Chronic Disease; Noncommunicable Diseases | interventions — Tacrine

STUDY DESIGN:
Intervention Model Description: Single-arm quasi-experimental study for evaluating the effectiveness of a digital health program in weight reduction for the prevention of non-communicable diseases in the Thai workplace setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Intervention Arm (Experimental): Participants will engage in various activities, including:
  * Attending four group health education sessions, each lasting one hour, over a six-month period.
  * Having access to individual chat consultations with a healthcare team, including doctors, dietitians, fitness coaches, and psychologists, available from 9:00 AM to 5:00 PM on workdays, excluding public holidays, with no limit on consultation times.
  Interventions: Behavioral: A Digital Health Program for Non-Communicable Disease Prevention in a Workplace Setting in Thailand

INTERVENTIONS:
Behavioral: A Digital Health Program for Non-Communicable Disease Prevention in a Workplace Setting in Thailand — The program consists of two main components: (1) Participants are invited to join health courses and/or health activities in the form of seminars or group activities, and (2) Participants will have access to an application that is part of the program, where they can consult with health experts to plan lifestyle modifications and reduce behavioral risk factors over the 6-month duration of the research project, totaling four sessions, each lasting one hour.

SUMMARY:
The goal of this quasi-experimental study is to test the effectiveness of a digital health program designed to prevent non-communicable diseases (NCDs) in employees within a workplace setting in Thailand. The main questions it aims to answer are:

* Can a digital health program help participants lose weight?
* Does the digital health program improve other health outcomes such as Body Mass Index (BMI), blood lipid levels (triglycerides and LDL), blood sugar levels (HbA1c or fasting plasma glucose), and blood pressure? Is the digital health program feasible and acceptable in the Thai workplace setting, as measured by participation rates, usage, and participant satisfaction?

Participants will:

* Attend four group health education sessions, each lasting one hour, scheduled over a six-month period.
* Have unlimited access to individual chat consultations with a healthcare team, including doctors, dietitians, fitness coaches, and psychologists, available from 9:00 AM to 5:00 PM on workdays, excluding public holidays.

DETAILED DESCRIPTION:
This quasi-experimental study titled "A Digital Health Program for Non-Communicable Disease Prevention in a Workplace Setting in Thailand" aims to evaluate the preliminary effectiveness of a digital health program in reducing weight among participants in a workplace setting. Conducted at Chulalongkorn Hospital, Bangkok, over a period of 1.5 years, the study focuses on the impact of the digital health program on various health outcomes, including Body Mass Index (BMI), blood lipid levels (triglycerides and LDL), blood sugar levels (HbA1c or fasting plasma glucose), and blood pressure. Additionally, it assesses the feasibility and acceptability of the program within the Thai workplace context, measured by participation rates, usage, and participant satisfaction.

The research adopts a single-arm quasi-experimental design to assess the weight loss efficacy of the digital health program aimed at preventing non-communicable diseases (NCDs) among employees at risk. The target population includes employees of the Faculty of Medicine, Chulalongkorn University, and/or Chulalongkorn Hospital, with an estimated sample size of 150 participants. Recruitment leverages employee health examination data, with informed consent obtained through comprehensive information sharing.

The intervention comprises four group health education sessions (1 hour each) and unlimited individual chat consultations during work hours, facilitated by a multidisciplinary team including doctors, dietitians, fitness coaches, and psychologists. Data collection spans six months, with a follow-up health examination at the six-month mark, coordinated by the Department of Preventive and Social Medicine, Chulalongkorn Hospital.

The research study conducted a series of educational sessions over six months, focusing on health goal setting, nutrition, physical fitness, psychological resilience, and health outcome evaluation. Here's a summary of the sessions conducted:

Health Goal Setting Lecture (Month 1): Participants learned about the importance of understanding their health, covering basics such as motivation for change, health risk assessment, introduction to the program's curriculum, and setting personal health goals using a realistic behavioral goal-setting framework.

Nutrition Lecture by a Dietitian (Month 2): This session introduced participants to creating a personalized eating plan and understanding individual nutrition. It explored topics like portion control and food selection, illustrated with successful case examples to demonstrate effective dietary strategies. The session concluded with the creation of a customizable eating plan and ongoing support through chat throughout the program.

Fitness Coaching Lecture (Month 3): A fitness coach introduced the appropriate amount, timing, and types of exercise, using successful case examples to show how to implement a real-life exercise plan. This laid the foundation for exercise plans aligned with health goals and encouraged participation in physical activities. The session ended with the creation of a tailored exercise plan and continuous modification support via chat throughout the program.

Psychology Lecture by a psychologist (Months 4-5): The session provided knowledge on coping plans for when goals are not met as intended, encouraging participants to develop their own coping strategies and build resilience. The importance of social support and resilience in maintaining healthy physical activities and eating habits to prevent reverting to old behaviors was emphasized. Participants were advised to review their health goals and received feedback on their physical and dietary practices.

Health Outcome Evaluation by a Doctor (Month 6): Participants met with a doctor for a scheduled physical examination six months after joining the research program. This included blood tests (6-12 milliliters, approximately 2 teaspoons) to assess laboratory results such as weight, Body Mass Index (BMI), lipid levels, blood sugar levels, and blood pressure.

All activities and processes are conducted remotely, utilizing digital platforms for both individual consultations and group training sessions. The study plans to tailor interventions to individual participants based on the Health Action Process Approach (HAPA), aiming for personalized behavior change support. Modifications to the trial, if any, will be documented upon completion. The trial's effectiveness and participant adherence will be assessed and recorded, ensuring a consistent approach throughout the program and documenting all digital platform interactions.

ELIGIBILITY:
Inclusion Criteria:

* Must have a Body Mass Index (BMI) indicating overweight, specifically between 23.0 and 27.5 kg/m². OR
* Must have blood lipid levels indicating risk, such as triglyceride levels between 150 and 199 mg/dL or LDL levels between 160 and 189 mg/dL. OR
* Must have blood sugar levels indicating a pre-diabetic state, such as an HbA1c level between 5.7% and 6.4% or fasting plasma glucose levels between 100 and 125 mg/dL. OR
* Must have systolic blood pressure between 120 and 139 mmHg and/or diastolic blood pressure between 80 and 89 mmHg.
* Must be able to read and communicate in Thai to participate in project activities.
* Must have access to digital devices compatible with the digital health program, such as smartphones with operating systems equivalent to or higher than iOS 11 or Android 5.1, or computers capable of joining online seminars.
* Must consent to participate in the research study.

Exclusion Criteria:

* Pregnancy, bedridden state, or disability that limits mobility or the ability to exercise.
* History of non-communicable diseases, such as heart disease, stroke, diabetes, or any acute illness.
* Participation in a health program or weight loss program currently or in the previous month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Weight | 6 months
  To assess weight reduction.

SECONDARY OUTCOMES:
BMI | 6 months
  To assess BMI change.
Total cholesterol | 6 months
  To assess total cholesterol change.
Triglycerides | 6 months
  To assess triglycerides change.
HDL | 6 months
  To assess HDL change.
LDL | 6 months
  To assess LDL change.
HbA1c | 6 months
  To assess HbA1c change.
Fasting plasma glucose | 6 months
  To assess fasting plasma glucose change.
blood pressure | 6 months
  To assess blood pressure change.
Feasibility (number of consented participants to all eligible participants ratio) | 3 months (recruitment period)
  number of consented participants to all eligible participants ratio
Acceptability | 6 months
  Net Promoter Score assessed by 1 verbal question at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jate Ratanachina, MD MSc PhD, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] กลุ่มเทคโนโลยี ระบาดวิทยา และมาตรการชุมชน กองโรคไม่ติดต่อ กรมควบคุมโรค กระทรวงสาธารณสุข. รายงานสถานการณ์โรค NCDs เบาหวาน ความดันโลหิตสูง และปัจจัยเสี่ยงที่เกี่ยวข้อง. 2020.
- [Background] คณะกรรมการเศรษฐกิจและสังคมแห่งเอเชียและแปซิฟิก. เหตุผลสนับสนุนการลงทุนใน มาตรการป้องกันและควบคุมโรคไม่ติดต่อในประเทศไทย. 2021.
- [Background] มูลนิธิสถาบันวิจัยและพัฒนาผู้สูงอายุไทย. สถานการณ์ผู้สูงอายุไทย พ.ศ. 2564. 2021.
- [Background] World Health Organization. Noncommunicable diseases. Fact sheets 2023 16 September 2023 [cited 2023 16 November 2023]; Available from: https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases.
- [Background] Burton, J. WHO healthy workplace framework and model: background and supporting literature and practices. 2010: Geneva.
- [Background] World Health Organization. World mental health report: transforming mental health for all. 2022: Geneva.
- [Background] World Health Organization. The impact of the COVID-19 pandemic on noncommunicable disease resources and services: results of a rapid assessment. 2020.
- [Background] วารณี บุญช่วยเหลือ, ทิพาพร พงษ์เมษา, และ กมลภัทร ไชยกิตติโสภน. การดําเนินงานลดเสี่ยงต่อโรคหัวใจและหลอดเลือดในกลุ่มวัยทํางาน ที่มีความคุ้มค่าหรือมีประสิทธิผล ในชุมชน สถานบริการสุขภาพและสถานที่ทํางาน. 2018.
- [Background] World Health Organization. Global Strategy on Diet, Physical Activity and Health. 2004, World Health Organization: Global Strategy on Diet, Physical Activity and Health.
- [Background] World Health Organization. Preventing Non Communicable Diseases in the Workplace through Diet and Physical Activity. 2008, World Health Organization, Geneva: WHO/World Economic Forum Report of a Joint Event.
- [Background] Proper KI, van Oostrom SH. The effectiveness of workplace health promotion interventions on physical and mental health outcomes - a systematic review of reviews. Scand J Work Environ Health. 2019 Nov 1;45(6):546-559. doi: 10.5271/sjweh.3833. Epub 2019 May 28. PMID 31134284
- [Background] Hafez D, Fedewa A, Moran M, O'Brien M, Ackermann R, Kullgren JT. Workplace Interventions to Prevent Type 2 Diabetes Mellitus: a Narrative Review. Curr Diab Rep. 2017 Feb;17(2):9. doi: 10.1007/s11892-017-0840-0. PMID 28150162
- [Background] Schwarz PEH, Timpel P, Harst L, Greaves CJ, Ali MK, Lambert J, Weber MB, Almedawar MM, Morawietz H. Blood Sugar Regulation for Cardiovascular Health Promotion and Disease Prevention: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Oct 9;72(15):1829-1844. doi: 10.1016/j.jacc.2018.07.081. PMID 30286928
- [Background] Cannon MJ, Ng BP, Lloyd K, Reynolds J, Ely EK. Delivering the National Diabetes Prevention Program: Assessment of Enrollment in In-Person and Virtual Organizations. J Diabetes Res. 2022 Feb 1;2022:2942918. doi: 10.1155/2022/2942918. eCollection 2022. PMID 35118160
- [Background] Moungngern Y, S.S., Teparak P, Sriwijitkamol A. Effects of a Health Promotion Program Conducted by Nurses on Stabilization of HbA1C in Subjects at Risk for Diabetes: A Phase III Randomized Controlled Trial. J Med Assoc Thai, 2018. 101(10): p. 1343-8.
- [Background] Dunkley AJ, Bodicoat DH, Greaves CJ, Russell C, Yates T, Davies MJ, Khunti K. Diabetes prevention in the real world: effectiveness of pragmatic lifestyle interventions for the prevention of type 2 diabetes and of the impact of adherence to guideline recommendations: a systematic review and meta-analysis. Diabetes Care. 2014 Apr;37(4):922-33. doi: 10.2337/dc13-2195. PMID 24652723
- [Background] Van Rhoon L, Byrne M, Morrissey E, Murphy J, McSharry J. A systematic review of the behaviour change techniques and digital features in technology-driven type 2 diabetes prevention interventions. Digit Health. 2020 Mar 24;6:2055207620914427. doi: 10.1177/2055207620914427. eCollection 2020 Jan-Dec. PMID 32269830
- [Background] World Health Organization. Self-care interventions for health. Self-care interventions for health 2022 [cited 2023 19 November 2023]; Available from: https://www.who.int/news-room/fact-sheets/detail/self-care-health-interventions.
- [Background] Skinner, D., S. Pete, and E.-O. Austen. Self-Care 2030: What does the future for health & wellbeing look like & how do we get there?, in School of Public Health. 2023.
- [Background] Zhang CQ, Zhang R, Schwarzer R, Hagger MS. A meta-analysis of the health action process approach. Health Psychol. 2019 Jul;38(7):623-637. doi: 10.1037/hea0000728. Epub 2019 Apr 11. PMID 30973747
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Schwarzer, R. Modeling Health Behavior Change: How to Predict and Modify the Adoption and Maintenance of Health Behaviors. Applied Psychology, 2008. 57(1): p. 1-29.
- [Background] Schwarzer, R. Health action process approach (HAPA) as a theoretical framework to understand behavior change. Actualidades en Psicología, 2016. 30(121): p. 119-130.
- [Result] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Result] Katula JA, Dressler EV, Kittel CA, Harvin LN, Almeida FA, Wilson KE, Michaud TL, Porter GC, Brito FA, Goessl CL, Jasik CB, Sweet CMC, Schwab R, Estabrooks PA. Effects of a Digital Diabetes Prevention Program: An RCT. Am J Prev Med. 2022 Apr;62(4):567-577. doi: 10.1016/j.amepre.2021.10.023. Epub 2022 Feb 10. PMID 35151522
- [Result] Aekplakorn W, Tantayotai V, Numsangkul S, Tatsato N, Luckanajantachote P, Himathongkam T. Evaluation of a Community-Based Diabetes Prevention Program in Thailand: A Cluster Randomized Controlled Trial. J Prim Care Community Health. 2019 Jan-Dec;10:2150132719847374. doi: 10.1177/2150132719847374. PMID 31079517